CLINICAL TRIAL: NCT07262658
Title: Disparities in Neurocognitive Impairment Among Hispanics/Latinos in the US With Parkinson's Disease: The Role of Cardiovascular Risk
Brief Title: Cognitive Disparities in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00115158; 801968 (Other: UC San Diego); Pro00115158 (Other: Duke University Health System)
Record Dates: First submitted 2023-08-08; First posted 2025-12-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hispanics with Parkinson's Disease: All Hispanics with PD will complete comprehensive neuromedical and neuropsychological evaluations, a blood draw and assessments of socio-cultural factors (e.g., health literacy, access to care, acculturation, bilingualism, discrimination, socioeconomic status).
  Interventions: Other: Will examine how Cardiovascular Disease risk, PD severity and social determinants impact neurocognitive impairment in Hispanics vs non-Hispanics Whites
- non-Hispanic Whites with Parkinson's Disease: All non-Hispanic Whites with PD will complete comprehensive neuromedical and neuropsychological evaluations, a blood draw and assessments of socio-cultural factors (e.g., health literacy, access to care, acculturation, bilingualism, discrimination, socioeconomic status).
  Interventions: Other: Will examine how Cardiovascular Disease risk, PD severity and social determinants impact neurocognitive impairment in Hispanics vs non-Hispanics Whites

INTERVENTIONS:
Other: Will examine how Cardiovascular Disease risk, PD severity and social determinants impact neurocognitive impairment in Hispanics vs non-Hispanics Whites — All participants will complete comprehensive neuromedical and neuropsychological evaluations, a blood draw and assessments of socio-cultural factors (e.g., health literacy, access to care, acculturation, bilingualism, discrimination, socioeconomic status).

SUMMARY:
This study will investigate disparities in neurocognitive impairment (NCI) among Hispanics/Latinos/as/x (henceforth Hispanics) living in the US-Mexico borderland of California or in North Carolina with Parkinson's Disease (PD) and determine mechanisms underlying these disparities. NCI is an important aspect of the clinical course of PD, particularly among Hispanics, who have increased prevalence of dementia. Among the many potential factors driving this disparity, the investigators chose to focus on a modifiable risk factor to which Hispanics are particularly vulnerable, and that has been linked to increased NCI, namely cardiovascular (CVD) risk (e.g., diabetes, hypertension, obesity).

DETAILED DESCRIPTION:
The proposed study will use a cross-sectional design to determine the presence of NCI in 120 persons with PD (age 40+), living in the US-Mexico borderland of California or in North Carolina, including 60 Hispanics and 60 non-Hispanic Whites. All participants will complete comprehensive neuromedical and neuropsychological evaluations, a blood draw and assessments of socio-cultural factors (e.g., health literacy, access to care, acculturation, bilingualism, discrimination, socioeconomic status). Using these data we will examine the extent to which CVD risk (e.g., diabetes, hypertension, obesity), PD severity and social determinants of health drive NCI among Hispanics with PD. The present proposal will capitalize on the infrastructure and expertise available at Duke University and will follow a community-based participatory research approach to complete the proposed study aims.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old and older
* non-Hispanic Whites
* Hispanics
* All genders
* Ability to provide consent
* Diagnosed with Parkinson's Disease

Exclusion Criteria:

* Other neurological illness/diagnosis
* Injury that would affect cognition (i.e. stroke, closed head injury with loss of consciousness for longer than 30 minutes)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed study will use a cross-sectional design to determine the presence of NCI in 120 persons with PD (age 40+), including 60 Hispanics and 60 non-Hispanic Whites living in the US/Mexico borderland of California or in North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Language (Letter Fluency) | Day 1 (day of enrollment)
Language (Animal Fluency) | Day 1 (day of enrollment)
Language (Vegetable Fluency) | Day 1 (day of enrollment)
Language (Multilingual Naming Test) | Day 1 (day of enrollment)
Speed of Information Processing | Day 1 (day of enrollment)
  Trail Making Test A
Speed of Information Processing | Day 1 (day of enrollment)
  WAIS-III Digit Symbol
Speed of Information Processing | Day 1 (day of enrollment)
  WAIS-III Symbol Search (Wechsler Adult Intelligence Scale)
Attention/Working Memory | Day 1 (day of enrollment)
  PASAT-50 (Paced Auditory Serial Addition Test)
Attention/Working Memory | Day 1 (day of enrollment)
  Number Span
Executive Function | Day 1 (day of enrollment)
  Trail Making Test B
Executive Function | Day 1 (day of enrollment)
  WCST-64 (Wisconsin Card Sorting Test)
Verbal Learning and Memory | Day 1 (day of enrollment)
  Hopkins Verbal Learning Test-Revised
Verbal Learning and Memory | Day 1 (day of enrollment)
  Craft Story Learning & Recall
Visual Learning and Memory | Day 1 (day of enrollment)
  Brief Visuospatial Memory Test - Revised, Benson Figure Delay
Visual-Spatial skills | Day 1 (day of enrollment)
  Benson Figure Copy
Everyday Functioning | Day 1 (day of enrollment)
  Modified Lawton-Brody Instrumental Activities of Daily Living questionnaire
Diagnosis of MCI/dementia in PD | Day 1 (day of enrollment)
  Objective presence of MCI and dementia in PD will be determined via comprehensive diagnostic criteria
diabetes mellitus | Day 1 (day of enrollment)
  fasting plasma glucose >126 mg/dL, an HbA1c >6.5%, or use of antihyperglycemic medications
hypercholesterolemia and dyslipidemia | Day 1 (day of enrollment)
  total cholesterol >240 mg/dL, LDL cholesterol >160 mg/dL, or HDL cholesterol <40 mg/dL or on cholesterol-lowering medication
hypertension | Day 1 (day of enrollment)
  systolic blood pressure >140 mm Hg, diastolic blood pressure >90 mm Hg, or on antihypertensive medication
current cigarette smoking | Day 1 (day of enrollment)
  Self-report
obesity | Day 1 (day of enrollment)
  BMI of >30.0
Parkinson's disease severity | Day 1 (day of enrollment)
  Movement Disorders Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Marquine, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - UC San Diego, La Jolla, California
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
Study is conducted only at these sites, hence there is no need to share information with other investigators.

REFERENCES:
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Background] Marquine MJ, Rivera Mindt M, Umlauf A, Suarez P, Kamalyan L, Morlett Paredes A, Yassai-Gonzalez D, Scott TM, Heaton A, Diaz-Santos M, Gooding A, Artiola I Fortuny L, Heaton RK, Cherner M. Introduction to the Neuropsychological Norms for the US-Mexico Border Region in Spanish (NP-NUMBRS) Project. Clin Neuropsychol. 2021 Feb;35(2):227-235. doi: 10.1080/13854046.2020.1751882. Epub 2020 May 20. PMID 32431209
- See also: recruitment flyer - Spanish — https://neurosciences.ucsd.edu/centers-programs/movement-disorders/research/801968-Neurocog-Flyer-SPANISH-06-Jun-2023-UCSD-IRB-Approved.pdf
- See also: recruitment flyer - English — https://neurosciences.ucsd.edu/centers-programs/movement-disorders/research/801968-Neurocog-Flyer-ENGLISH.pdf
- See also: Research Studies - Parkinson's Disease — https://neurosciences.ucsd.edu/centers-programs/movement-disorders/research/pd-studies.html